CLINICAL TRIAL: NCT02519127
Title: Employing Dynamic Kinetic Responses to Demonstrate the Effectiveness of Dietary Intervention: A Challenge-based Study Using a Low-glycaemic Load Diet
Brief Title: Metflex: The Effectiveness of a Dietary Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: NL52245.068.15/METC153004
Record Dates: First submitted 2015-07-07; First posted 2015-08-10 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Metabolic Flexibility
MeSH Terms: interventions — Diet, Western

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low glycaemic load diet (Experimental): Subjects will be following a low glycaemic load diet, typically high in polyphenols, proteins, vegetables, pulses, fibres and nuts, and low in glycemic carbohydrates, for six continuous weeks.
  Interventions: Other: Low glycaemic load diet
- Western diet (Experimental): Subjects will be following a western diet, typically high in saturated fat, refined sugars and salt, and low in fruit and vegetables and fibers, for six continuous weeks.
  Interventions: Other: Western diet

INTERVENTIONS:
Other: Low glycaemic load diet — Subjects will first be subjected to a 2-week run-in diet consisting of products that fit into a typical 'Western' diet. Thereafter subjects will be allocated to a low glycemic load diet for 6 weeks.
  Arms: Low glycaemic load diet
Other: Western diet — Subjects will first be subjected to a 2-week run-in diet consisting of products that fit into a typical 'Western' diet. Thereafter subjects will be allocated to a 'Western' diet for 6 weeks.
  Arms: Western diet

SUMMARY:
This study is testing the effectiveness of a dietary intervention by means of measuring the change in RQ upon a hyperinsulinemic euglycemic clamp challenge and by means of measuring the kinetic responses of multiple PF markers (including RQ) to an acute mixed meal challenge before and after a 6-week dietary intervention. The challenges will be applied to investigate whether the kinetic response is a better measure for health and wellbeing when compared to fasting (baseline) levels. In addition, several measures that reflect perceivable benefits like mood, quality of life, sleep quality, cognitive and physical performance will be assessed in a first exploratory attempt to link (changes in) PF to consumer perceivable benefits.

Subjects will be randomly allocated to a low glycemic load diet or a 'Western' diet for 6 weeks. Before and after the intervention several measurements will take place. The low glycemic load diet will be high in polyphenols, protein, vegetables, pulses, fibres and nuts, and low in glycemic carbohydrates. All these dietary factors have been shown to improve glycemic control and/or to reduce metabolic syndrome risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Men and postmenopausal women: ≥ 50 and ≤ 70 years at the start of the study
* Body mass index (BMI) ≥ 25.0 and ≤ 35.0 kg/m2
* Healthy (as determined by dependent physician): no medical conditions which might affect the study measurements, absorption, metabolism and distribution (including diabetes type 1 and type 2, gastrointestinal dysfunction, gastrointestinal surgery and inflammatory diseases) as assessed by physical characteristics and health and lifestyle questionnaire
* Fasting blood glucose value ≤ 6.9 mmol/litre at screening
* Waist circumference >94 cm for males, >80 cm for females
* Maximum 2.5 hours of moderate to vigorous physical activity per week (during last 3 months)
* Agreeing to be informed about medically relevant personal test-results by a physician
* Willing to comply to study protocol during study
* Accessible veins on arms as determined by examination at screening

Exclusion Criteria:

* Reported participation in another nutritional or biomedical trial three months before the pre-study examination or during the study
* Blood donation in the past three months
* Reported participation in night shift work two weeks prior to pre-study investigation or during the study. Night work is defined as working between midnight and 6.00 AM;
* Consumption of > 21 alcoholic units for males, > 14 alcohol units for females in a typical week;
* Reported use of any nicotine containing products in the six months preceding the study and during the study itself;
* Reported dietary habits: medically prescribed diet, slimming diet, vegetarian;
* People who are familiar with an allergy or intolerance to any of the provided food products
* Reported weight loss or weight gain (10%) in the last six months prior to the pre-study screening;
* Clinically relevant abnormalities in clinical chemistry at screening (to be judged by the study physician);
* Being an employee of Unilever or the collaborating research departments in Maastricht University Medical Centre (MUMC+);
* Taking medication, which may interfere with study measurements, as judged by the responsible physician;
* Subjects, who do not want to be informed about unexpected medical findings, or do not wish that their treating physician is informed.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-07; Primary Completion 2017-05-12 (Actual); Study Completion 2017-05-12 (Actual)

PRIMARY OUTCOMES:
Metabolic flexibility, as measured by delta RQ (change in RQ) upon a hyperinsulinemic euglycemic clamp | Within 5 days before the start of the 6 week dietary intervention and again in the 6th week of the dietary intervention

SECONDARY OUTCOMES:
Metabolic flexibility, as measured by delta RQ (change in RQ) upon a mixed meal challenge | Within 5 days before the start of the 6 week dietary intervention and again in the 6th week of the dietary intervention
Phenotypic flexibility markers, as measured by various blood parameters such as lipids, glucose, inflammatory markers and more, upon a mixed meal challenge | Within 5 days before the start of the 6 week dietary intervention and again in the 6th week of the dietary intervention
Diet-induced changes in the Kinetic responses vs. the baseline values of RQ and various phenotypic flexibility parameters such as lipids, glucose, inflammatory markers and more | Within 5 days before the start of the 6 week dietary intervention and again in the 6th week of the dietary intervention
Phenotypic flexibility markers, as measured by various blood parameters such as lipids, glucose, inflammatory markers and more, in the fasted state | Within 5 days before the start of the 6 week dietary intervention and again in the 6th week of the dietary intervention
Insulin sensitivity, as measured by a hyperinsulinemic euglycemic clamp | Within 5 days before the start of the 6 week dietary intervention and again in the 6th week of the dietary intervention

OTHER OUTCOMES:
Functional markers of cognitive performance, as measured by attention, memory and executive function | Within 5 days before the start of the 6 week dietary intervention and again in the 6th week of the dietary intervention
Functional markers of physical performance, as measured by the timed up-and-go test (TUGT), the 6-minute walk test, handgrip and muscle strength tests | Within 5 days before the start of the 6 week dietary intervention and again in the 6th week of the dietary intervention
Sleep quality, as assessed with the10-item Pittsburgh Sleep Quality Index | Within 5 days before the start of the 6 week dietary intervention and again in the 6th week of the dietary intervention
Mood, as assessed by the Affect grid | Within 5 days before the start of the 6 week dietary intervention and again in the 6th week of the dietary intervention
Quality of life, as assessed by a 32-item questionnaire, including social, spiritual, emotional, cognitive, physical, activities of daily living and integrated quality of life | Within 5 days before the start of the 6 week dietary intervention and again in the 6th week of the dietary intervention
Body composition, as measured by the deuterium water method | Within 5 days before the start of the 6 week dietary intervention and again in the 6th week of the dietary intervention
36-hour blood pressure, as measured by the continuous blood pressure device mobil-o-graph | 36 hours within 5 days before the 6 week dietary intervention and again 36 hours in the 6th week of the dietary intervention
36-hour glycaemic response, as measured by the continuous blood glucose device ipro2 (Medtronic) | 36 hours within 5 days before the 6 week dietary intervention and again 36 hours in the 6th week of the dietary intervention

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schrauwen, Professor, Principal Investigator — Maastricht University Medical Center; Ronald Mensink, Professor, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

REFERENCES:
- [Derived] Fechner E, Bilet L, Peters HPF, Schrauwen P, Mensink RP. A Whole-Diet Approach Affects Not Only Fasting but Also Postprandial Cardiometabolic Risk Markers in Overweight and Obese Adults: A Randomized Controlled Trial. J Nutr. 2020 Nov 19;150(11):2942-2949. doi: 10.1093/jn/nxaa252. PMID 33096554
- [Derived] Fechner E, Bilet L, Peters HPF, Hiemstra H, Jacobs DM, Op 't Eyndt C, Kornips E, Mensink RP, Schrauwen P. Effects of a whole diet approach on metabolic flexibility, insulin sensitivity and postprandial glucose responses in overweight and obese adults - A randomized controlled trial. Clin Nutr. 2020 Sep;39(9):2734-2742. doi: 10.1016/j.clnu.2019.12.010. Epub 2019 Dec 17. PMID 31899037